CLINICAL TRIAL: NCT06090812
Title: Initial Volume Status in Patients With Acute Brain Injury is Associated With Neurological Prognosis
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-PUMCH-A-266
Record Dates: First submitted 2023-10-14; First posted 2023-10-19 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2023-10

CONDITIONS: Acute Brain Injury; Paroxysmal Sympathetic Hyperactivity; Volume Status; Right Heart Function; Right Cardiogenic Pulmonary Edema; Glasgow Outcome Scale Extended
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- acute brain injury: The included population was patients with acute brain injury, protected from acute cerebrovascular events, traumatic brain injury, and acute cerebral edema. Assessment of stress levels, Ultrasound evaluation of volume status, right heart function, and pulmonary edema.
  Interventions: Other: Ultrasound evaluation

INTERVENTIONS:
Other: Ultrasound evaluation — Ultrasound evaluation of volume status, right heart function, and pulmonary edema.

SUMMARY:
In this study, we investigated the clinical variability in paroxysmal sympathetic hyperactivity in patients with acute brain injury and examined the prognostic value of the Paroxysmal Sympathetic Hyperactivity Assessment Measure (PSH-AM) in relation to Doppler ultrasound assessment of volume status, right heart function, and pulmonary edema. Thirty patients with ABI were prospectively enrolled. A correlation analysis between the PSH-AM score and related clinical indicators was performed using Pearson's or Spearman's correlation coefficient. Receiver operating characteristic curves were used to assess the prediction of the 6-month Glasgow Outcome Scale Extended score for neurorehabilitation prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Only adult patients (>18 years of age) were included. The other inclusion criteria were 1) definite cerebrovascular accident or craniocerebral injury (a clear change in consciousness or suggestive imaging); 2) the ability to undergo ultrasound to obtain information on volume status and cardiac and pulmonary monitoring; and 3) fulfilment of the measurement conditions.

Exclusion Criteria:

* The exclusion criteria were 1) a history of cardiovascular disease, such as coronary artery disease, heart failure, or atrial fibrillation; 2) presence of severe valvular disease or an EF of <30%; 3) chronic lung disease; 4) chronic liver failure or renal insufficiency; 5) comorbid malignant neoplasm or acute/chronic infectious disease prior to craniocerebral injury; 6) pregnancy or breastfeeding; 7) history of psychiatric disorders; 8) history of drug abuse or alcohol misuse; 9) history of β-blocker use; 10) comorbid spinal cord injury; 11) death or discharge from hospital within 5 days of hospitalization.

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Only adult patients (>18 years of age) were included. The other inclusion criteria were a definite cerebrovascular accident or craniocerebral injury (a clear change in consciousness or suggestive imaging); the ability to undergo an ultrasound to obtain information on volume status and cardiac and pulmonary monitoring; and fulfillment of the measurement conditions.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Assessment of stress levels | Day 1, Day 3, Day 5
  The PSH-AM score is the sum of the CFS and DLT scores, and assesses the likelihood of a diagnosis of PSH. A score of <8 means that PSH is unlikely, 8-16 suggests that PSH is likely, and ≥17 suggests that PSH is highly likely.
Ultrasound evaluation of volume status | Day 1, Day 3, Day 5
  The cardiac ultrasound probe was placed under the xiphoid process, and the probe was moved from the upper abdominal position to the standard four-chamber view of the heart under the xiphoid process, where the right ventricle is first seen. The probe was rotated downward and toward the spine, with the directional marker pointing toward the patient's head, showing the inferior vena cava (IVC) entering the right atrium and the hepatic vein converging into the IVC. The IVC diameter was measured 2 cm from the entrance of the right atrium, and the ultrasound images were frozen at the end of expiration and at the end of inspiration to measure the maximum IVC diameter. Simultaneous measurement of central venous pressure (CVP) was obtained.
Ultrasound evaluation of right heart function | Day 1, Day 3, Day 5
  In the apical four-chamber view, a TDI sample volume was placed on the RV free wall at a distance of 1 cm from the tricuspid annulus.

CONTACTS AND LOCATIONS:
Locations (1):
- Wei Du, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No